CLINICAL TRIAL: NCT00043303
Title: A Multicenter Study of the Safety and Anti-Fibrotic Efficacy of Interferon-Gamma 1b (Actimmune) in Patients With Severe Lever Fibrosis or Compensated Cirrhosis Due to Hepatitis C.
Brief Title: Safety and Efficacy Study of Interferon Gamma-1b in Hepatitis C Patients With Liver Fibrosis or Cirrhosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: InterMune (Industry)
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GILF-001
Record Dates: First submitted 2002-08-07; First posted 2002-08-09 (Estimated); Last update posted 2007-11-01 (Estimated); Status verified 2007-10

CONDITIONS: Liver Fibrosis; Cirrhosis
Keywords: hepatitis C; liver fibrosis; liver cirrhosis
MeSH Terms: conditions — Liver Cirrhosis; Fibrosis; Hepatitis C | interventions — interferon gamma-1b

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: interferon gamma-1b — 100 or 200 mcg, SQ, 3x per week

SUMMARY:
The purpose of this research study is to test the safety and effectiveness of Interferon gamma-1b (IFN-g 1b) injected subcutaneously (under the skin) for the treatment of advanced liver fibrosis and cirrhosis in patients with chronic hepatitis C infections.

IFN-g 1b is not currently approved for the treatment of liver fibrosis.

DETAILED DESCRIPTION:
This study will evaluate the safety and tolerability of IFN-g 1b in patients with advanced liver fibrosis and cirrhosis due to hepatitis C. This study will also evaluate whether IFN-g 1b is effective in reducing the amount of fibrosis in the liver.

ELIGIBILITY:
* Men or women 18 to 75 years
* Chronic hepatitis C infection based on a history of positive anti-HCV antibody and/or HCV RNA
* History of prior treatment with interferon-a-based therapies or an assessment by the investigator that the patient would not benefit from interferon-a-based therapy or that treatment with interferon-a is contraindicated
* Stage 4, 5 or 6 liver fibrosis according to the Ishak scoring system.
* Cannot have presence of clinically evident ascites requiring active diuretic therapy, history of or therapy for hepatic encephalopathy, or history of GI variceal bleeding within the last 2 years (diuretic therapy of stable mild-to-moderate peripheral edema is permitted)
* Must meet minimum blood chemistry requirements
* Cannot have unstable or uncontrolled thyroid disease
* Cannot have a variety of other diseases (listed in protocol
* Other conditions for enrollment exist which would be discussed with a Clinician upon screening for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 502 (Actual)
Dates: Start 2001-09; Study Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
Ishak fibrosis score | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Steven Porter, MD, Study Director — InterMune